CLINICAL TRIAL: NCT07056764
Title: Development of Lung Vibration Equipment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burapha University (Other)
Responsible Party: Principal Investigator, Piyapong Prasertsri, Associate Professor Dr., Burapha University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB1-014/2568
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Sputum Removal

STUDY DESIGN:
Intervention Model Description: Patients who consent to participate in the study and pass the screening process will be randomly assigned by drawing lots to determine which type of lung vibration they will receive first. For all patients, lung vibration will be performed in conjunction with chest percussion and suctioning. Each volunteer will participate in the study for two days, receiving different treatments each day according to the randomly assigned order.
Masking Description: Masking will not be employed in this crossover study, as both participants and investigators will be aware of the intervention administered in each period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (Active Comparator): Patients who draw the standard lung vibration will receive manual chest vibration performed by a physical therapist for 1-2 minutes per time, continuously for at least 6 times per set, with a total duration not exceeding 30 minutes. On the following day, they will switch to the other procedure: lung vibration using the vibration device developed by the researcher, for 1-2 minutes per time, continuously for at least 6 times per set, with a total duration not exceeding 30 minutes as well (in conjunction with chest percussion and suctioning).
  Interventions: Other: Standard treatment
- Standard treatment + Lung vibration device (Experimental): Patients who draw the lung vibration using the vibration device will receive the procedure using the device developed by the researcher, for 1-2 minutes per time, continuously for at least 6 times per set, with a total duration not exceeding 30 minutes. On the following day, they will switch to the other procedure: standard manual lung vibration performed by a physical therapist, for 1-2 minutes per time, continuously for at least 6 times per set, with a total duration not exceeding 30 minutes as well (in conjunction with chest percussion and suctioning).
  Interventions: Device: Standard treatment + Lung vibration device

INTERVENTIONS:
Other: Standard treatment — Patients will be randomly assigned by drawing lots to determine the initial type of lung vibration treatment they will receive: either standard treatment alone or standard treatment combined with the lung vibration device.
  Arms: Standard treatment
Device: Standard treatment + Lung vibration device — Patients will be randomly assigned by drawing lots to determine the initial type of lung vibration treatment they will receive: either standard treatment alone or standard treatment combined with the lung vibration device.
  Arms: Standard treatment + Lung vibration device

SUMMARY:
This study designed a portable and easily accessible lung vibration device that is simple to use and can operate with both a battery system and a charging system for greater convenience. It helps enhance the effectiveness of mucus drainage, prevents complications, and reduces both the duration and cost of hospital treatment.

DETAILED DESCRIPTION:
Lung vibration device uses a motor as the power source to generate vibrations and has a shape similar to an iron. It is connected by an electrical cord in this section and can operate using either a battery system or a charging system. It features a vertically aligned handle perpendicular to the main body for a firm grip. The base of the device has a sponge head to absorb shock from the vibration during use, which is removable. The on/off switch is located at the end of the handle. This device uses 220-volt alternating current. The unit weighs approximately 1.1 kilograms and is made of strong and durable plastic.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-59 years
* Inpatients at Burapha University Hospital, Mueang District, Chonburi Province, with pulmonary secretion retention
* Referred by their attending physician for enhanced secretion clearance through physical therapy methods

Exclusion Criteria:

* Having inflamed wounds on the chest or back
* Having unstable vital signs, defined as: resting heart rate <60 or >100 beats per minute; blood pressure <90/60 or >120/80 mmHg; respiratory rate <12 or >20 breaths per minute; oxygen saturation <95%; and body temperature >37°C
* Having a bleeding tendency, defined as a platelet count <20,000 per cubic millimeter
* Taking medications that increase bleeding risk within 7 days prior to participation, including: Anticoagulants (such as Warfarin, Dabigatran, Rivaroxaban, Apixaban, Edoxaban), Antiplatelet agents (such as Aspirin, Clopidogrel, Dipyridamole, Prasugrel, Ticagrelor)
* Having an International Normalized Ratio (INR) >1.1 for those not on anticoagulants, and >3.0 for those on anticoagulants
* Having subcutaneous emphysema
* Experiencing severe hemoptysis (coughing up blood)
* Having chest wall pain
* Having acute spinal cord injury, rib fractures, or conditions associated with high fracture risk
* Having skin grafts or burn wounds
* Being admitted to intensive care units (ICU, RICU, or CICU)
* Having untreated pneumothorax
* Having an acute inflammatory process of the respiratory system
* Having inflammatory or infectious conditions such as tuberculosis, lung abscess, or COVID-19
* Having respiratory diseases that are contraindications or precautions for lung vibration, including COPD, uncomplicated pneumonia, asthma, lung cancer, or metastatic cancer

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2025-02-08 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | Baseline (0 minutes) and immediately post-intervention (30 minutes)
  Systolic blood pressure will be measured in mmHg unit
Diastolic blood pressure | Baseline (0 minutes) and immediately post-intervention (30 minutes)
  Diastolic blood pressure will be measured in mmHg unit
Body temperature | Baseline (0 minutes) and immediately post-intervention (30 minutes)
  Body temperature will be measured in degree Celsius
Oxygen saturation | Baseline (0 minutes) and immediately post-intervention (30 minutes)
  Partial pressure of oxygen saturation will be measured in percent
Sputum | Immediately post-intervention (30 minutes)
  Sputum will be measured for its quantity in ml unit and quality using photograph

CONTACTS AND LOCATIONS:
Overall Officials: Piyapong Prasertsri, Ph.D., Principal Investigator — Faculty of Allied Health Sciences, Burapha University
Locations (1):
- Burapha University Hospital, Mueang, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.